CLINICAL TRIAL: NCT07067840
Title: Safety and Efficacy of the Triple Branched Covered Stent Graft System for the Treatment of Aortic Arch Lesions: a Prospective, Multicenter, Single-Arm Trial.
Brief Title: Triple Branched Stent Graft System for Aortic Arch Lesions
Acronym: TRACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Zhongnan Hospital (Other); The University of HongKong-Shenzhen Hospital (Unknown); West China Hospital (Other); Meizhou People's Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The Third Affiliated Hospital of Wenzhou Medical University (Other); The First Affiliated Hospital of University of South China (Other); First Affiliated Hospital of Chongqing Medical University (Other); Guangyuan Central Hospital (Unknown); Jining First People's Hospital (Other); First People's Hospital of Yunnan Province (Unknown); Dalian Municipal Central Hospital (Other); Tianjin Chest Hospital (Other); Xiangya Hospital of Central South University (Other); The Affiliated Hospital Of Southwest Medical University (Other); Kunming Yan'an Hospital (Unknown)
Responsible Party: Principal Investigator, Qingsheng Lu, Dr., Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRACE-1
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Aortic Arch Aneurysm; Aortic Arch Pseudoaneurysm; Aortic Arch Ulcer
Keywords: triple branched stent graft; aortic arch; aortic ulcer; aortic aneurysm
MeSH Terms: conditions — Aneurysm, Aortic Arch; Aortic Aneurysm | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated with the triple branched stent graft system (Experimental): Participant group that treated with the triple branched stent graft system
  Interventions: Device: Treated with the triple branched stent graft system

INTERVENTIONS:
Device: Treated with the triple branched stent graft system — Participants treated with the triple branched stent graft system

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of the Triple Branched Covered Stent Graft System in treating aortic arch lesions. The main questions it aims to answer are:

* Does the Triple Branched Covered Stent Graft System achieve a 12-month treatment success rate that meets or exceeds the predefined target value?
* What is the 30-day major adverse event (MAE) rate following the use of the Triple Branched Covered Stent Graft System?

Researchers will use a single-arm study design with predefined target values for the primary endpoints to assess the performance of the stent system.

Participants will:

* Undergo a comprehensive screening process to determine eligibility based on specific inclusion and exclusion criteria.
* Receive the Triple Branched Covered Stent Graft System implantation as part of the treatment for their aortic arch lesions.
* Attend follow-up visits at specified intervals (e.g., pre-discharge, 30 days post-surgery, 6 months, 12 months, and annually up to 5 years) for evaluations including imaging studies (CTA) and clinical assessments.
* Report any adverse events or changes in their health status during the follow-up period.

ELIGIBILITY:
* Inclusion Criteria：

  1. Patients aged 18-80 years.
  2. Diagnosed with aortic arch lesions that require treatment, including true aortic arch aneurysms, false aortic arch aneurysms, and aortic arch ulcers.
  3. The investigator determines that the subject is suitable for endovascular therapy.
  4. The subject understands the purpose of the trial, voluntarily agrees to participate, and is willing to undergo follow-up.
  5. Anatomical conditions:

     * Ascending aorta length ≥50 mm.
     * Ascending aorta diameter ≥26 mm and ≤46 mm.
     * Proximal landing zone length ≥20 mm.
     * Brachiocephalic artery diameter ≤19 mm and ≥9 mm, with a length ≥20 mm.
     * Left common carotid artery and left subclavian artery diameter ≤13 mm and ≥5 mm, with a left common carotid artery length ≥20 mm, and the distance from the left vertebral artery opening to the left subclavian artery opening on the aorta ≥20 mm.
  6. The investigator assesses the subject as a high-risk patient for open surgery or with significant contraindications to open surgery.
* Exclusion Criteria

  1. Pregnant or breastfeeding women.
  2. Patients diagnosed with connective tissue diseases related to the aorta (e.g., Marfan syndrome).
  3. Infectious aortic diseases or Takayasu arteritis.
  4. Patients who have undergone endovascular treatment of the ascending aorta or aortic arch.
  5. Patients with a known allergy to nickel-titanium alloy, contrast agents, or other relevant materials.
  6. Severe renal failure (creatinine levels more than twice the upper limit of normal; dialysis patients are excluded).
  7. Hematological abnormalities:

     * Leukopenia (WBC < 3×10⁹/L).
     * Anemia (Hb < 70 g/L).
     * Coagulation disorders: thrombocytopenia (PLT count < 50×10⁹/L).
  8. Heart transplant recipients.
  9. History of myocardial infarction or stroke within the past 3 months.
  10. Heart function class IV (NYHA classification).
  11. Active infections, such as bacteremia or sepsis.
  12. Patients with an expected survival of less than 12 months.
  13. Patients with aortic valve replacement with a mechanical valve that would interfere with the safe introduction of the trial device.
  14. Subjects participating in other drug or medical device clinical trials and have not yet completed the primary endpoints of those trials.
  15. Poor compliance, with an expectation of inability to attend follow-up visits.
  16. Other conditions deemed by the investigator as unsuitable for endovascular therapy, such as severe vascular stenosis, calcification, tortuosity, thrombosis, or inability to cooperate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
12-month Treatment Success Rate | 12 months postoperatively
  Definition: Treatment success at 12 months is defined as immediate technical success, with no device/aneurysm-related death or unplanned secondary intervention postoperatively, and no increase in the diameter of the treated aorta segment (aneurysm or ulcer lesion diameter increased by ≥5mm) due to type I/III endoleak on CTA imaging follow-up at 12 months.
30-day Major Adverse Event Rate | 30 days postoperatively
  Any of the following events occurring within 30 days: 1.All-cause death: Any death from any cause within 30 days. 2.Disabling stroke: Defined as a Modified Rankin Scale (MRS) score ≥2 due to neurological deficits, with an increase of at least one grade from baseline. 3.Persistent paraplegia: Defined as a spinal ischemia grade ≥3 according to the spinal ischemia grading system. 4.Renal failure: New-onset persistent renal failure with a creatinine increase of more than 50% above preoperative levels, requiring dialysis. 5.Myocardial infarction: Clinically diagnosed as a new acute myocardial infarction, or requiring Percutaneous Coronary Intervention (PCI) or Coronary Artery Bypass Grafting (CABG). 6.Respiratory failure: Intubation for more than 1 week during hospitalization.

SECONDARY OUTCOMES:
Immediate Technical Success Rate | Immediately after the surgery
  The main and branch stents are successfully delivered to the predetermined position, accurately positioned and successfully deployed, the main and branch delivery systems are safely removed from the body, there is no branch stent stenosis or occlusion, and no device/aneurysm-related death or unplanned additional surgery.
Branch Stent Patency Rate | pre-discharge, at 30 days, 6 months, 12 months, and annually at 2, 3, 4, and 5 years postoperatively
  Based on imaging follow-up using Digital Subtraction Angiography (DSA) or Computed Tomographic Angiography (CTA), the degree of stenosis in the branches of the brachiocephalic artery, left common carotid artery, and left subclavian artery is ≤50%.
All-cause Mortality Rate | pre-discharge, at 30 days, 6 months, 12 months, and annually at 2, 3, 4, and 5 years postoperatively
  The rate of death from any cause postoperatively.
Aortic Lesion-related Mortality Rate | pre-discharge, at 30 days, 6 months, 12 months, and annually at 2, 3, 4, and 5 years postoperatively
  The rate of death related to aortic lesions.
Paraplegia Incidence Rate | pre-discharge, at 30 days, 6 months, 12 months, and annually at 2, 3, 4, and 5 years postoperatively
  Assessed using the spinal ischemia grading system, with the grade recorded.
Stroke Incidence Rate | pre-discharge, at 30 days, 6 months, 12 months, and annually at 2, 3, 4, and 5 years postoperatively
  Assessed using the Modified Rankin Scale (MRS), with the grade recorded.
Secondary Intervention Incidence Rate | pre-discharge, at 30 days, 6 months, 12 months, and annually at 2, 3, 4, and 5 years postoperatively
  Includes open or endovascular surgery caused by type I/III endoleak, aortic growth (caused by type I/III endoleak), aortic rupture, branch stenosis or occlusion, stent migration, or new-onset dissection at the proximal or distal end, excluding planned expected surgery.
Stent Fracture/Twist/Collapse Incidence Rate | pre-discharge, at 30 days, 6 months, 12 months, and annually at 2, 3, 4, and 5 years postoperatively
  The incidence of stent fracture, twist, or collapse detected by imaging postoperatively.
Stent Migration Incidence Rate | pre-discharge, at 30 days, 6 months, 12 months, and annually at 2, 3, 4, and 5 years postoperatively
  The incidence of stent migration ≥10mm.
Endoleak Incidence Rate | pre-discharge, at 30 days, 6 months, 12 months, and annually at 2, 3, 4, and 5 years postoperatively
  Based on imaging results from DSA or CTA, the incidence of endoleak postoperatively. Endoleak is classified as follows: Type I refers to blood reflux at the proximal and distal ends of the stent; Type II refers to retrograde blood flow from the aortic branch vessels; Type III refers to blood reflux at the site of stent membrane rupture or stent connection; Type IV refers to leakage of the covered stent membrane.
Maximum Diameter and Diameter Change of Aortic Lesion | pre-discharge, at 30 days, 6 months, 12 months, and annually at 2, 3, 4, and 5 years postoperatively
  The maximum diameter of the aortic lesion segment is recorded preoperatively and during postoperative follow-up, measured perpendicular to the centerline. The proportions of maximum diameter reduction ≥5mm, maximum diameter increase ≥5mm, and maximum diameter change less than 5mm are calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Qingsheng Lu, Dr., Principal Investigator — Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Naval Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No